CLINICAL TRIAL: NCT02318472
Title: Effects of Direct Functional Mobilization After Achilles Tendon Rupture on Healing and Outcome
Brief Title: Early Mobilization After Achilles Tendon Rupture
Acronym: EarlyM-Achil
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: OPED GmbH (Unknown)
Responsible Party: Principal Investigator, Paul Ackermann, Associate Professor, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR2012-2510
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Achilles Tendon Rupture; Deep Venous Thrombosis
Keywords: Microdialysis; Patient related outcome; Heel rise test; Immobilization; functional mobilization; Ultrasound
MeSH Terms: conditions — Venous Thrombosis | interventions — Casts, Surgical

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early mobilization (Experimental): Functional mobilization initiated directly post-operative with a weight-bearing VACOped orthosis with adjustable range of motion of the ankle
  Interventions: Device: VACOped orthosis
- Immobilization (Active Comparator): Treatment as usual using plaster cast immobilization
  Interventions: Device: Plaster cast

INTERVENTIONS:
Device: VACOped orthosis — Weight-bearing orthosis with adjustable range of motion of the ankle
  Arms: Early mobilization
Device: Plaster cast — Lower limb plaster cast
  Arms: Immobilization

SUMMARY:
The purpose of this study is to determine whether early mobilization after Achilles tendon rupture can speed up healing, prevent development of venous thromboembolism and improve patient outcome.

DETAILED DESCRIPTION:
Patients with acute Achilles tendon rupture will be screened for eligibility at the Karolinska University Hospital and Södersjukhuset, Stockholm.

One hundred-fifty patients will be included and enrolled and assigned to the interventions either by a third party nurse or by a research nurse. Randomisation will be performed with use of computer-generated random numbers in permuted blocks of four, through an independent software specialist, and consecutively numbered, sealed, opaque envelopes opened after surgery and prior to treatment.

The patients will be randomized to undergo either treatment as usual using plaster cast treatment alone or direct post-operative functional mobilization with a weight-bearing orthosis with adjustable range of motion of the ankle.

The power calculation was based upon data from a recent study reporting a 50% rate of CDU-verified DVT after ATR surgery (Domeij-Arverud et a. 2015). We estimated early functional mobilization (EFM) to confer a 50% risk reduction. Sixty-three patients in each group were required to detect a difference of 25% in the incidence of DVT (two-sided type-I error rate = 5%; power = 80%). We decided to include 150 patients to counteract drop-outs. On recommendations from the ethical committee, a ratio of 2:1 was chosen, since our hypothesis was that the EFM group would perform better.

The endpoint of the first part of the study is tendon healing quantified at 2 weeks by microdialysis followed by quantification of markers for tendon repair. The sample size for the outcome in the microdialysis study was calculated on a difference of the glutamate metabolite of 12 µM between the two groups. For this power analysis, we used a glutamate standard difference of 15 µM resulting from a previous study. It was determined that a sample size of 25 patients per group would be necessary to detect the glutamate difference with 80% power when alpha was set equal to 5%. Anticipating that we would lose 10% of participants enrolled, we plan to enroll 27 patients in each group for microdialysis.

The primary aim of the short-term follow up of this randomized, controlled trial was to assess the efficacy of EFM to reduce the DVT incidence after ATR surgery, at two and six weeks post-operatively, compared to treatment-as-usual, i.e. two weeks of plaster cast followed by four weeks' orthosis immobilization. The secondary aim was to evaluate the effect of patient intrinsic factors (age, BMI, calf circumference, ankle range of motion, pain and fear of movement) and patient extrinsic factors (amount of weightbearing, number of daily steps) on the risk of sustaining a DVT.

The primary aim with the long-term follow up is to investigate the effect of early postoperative functional mobilization compared to immobilization on patient-reported function, health, fear of movement, physical activity level, and differences in functional capacity. The second aim is to explore if the occurrence of DVT postoperatively effects functional outcome in the long-term after surgical treatment of ATR.

Additional aims:

The primary aim of the second part of this study was to assess the number of steps and the amount of loading in a weight bearing orthosis during the first six weeks post-surgical ATR repair. A secondary purpose was to investigate if the amount of loading was correlated to fear of movement or/and pain.

The aim with this substudy is to describe differences between the two groups over time regarding tendon elongation, differences in muscle cross-sectional area and differences in tendon cross-sectional area (on the injured side) and to examine if the differences can predict functional outcome in the long-term and if any of the follow-up occasions are most important for long-term functional outcome.

Few studies have evaluated outcome more than one year after injury. The aim of this substudy is to investigate differences in outcome at 3 years after injury between the patients that sustained a DVT and those who did not sustain a DVT. Another aim is to compare the two intervention groups over 3-years time.

ELIGIBILITY:
Inclusion Criteria:

* Acute unilateral ATR, operated on within 96 hours
* Age between 18 and 75 years

Exclusion Criteria:

* Inability to give informed consent
* Current anticoagulation treatment (including high dose acetylsalicylic acid)
* Planned follow-up at other hospital
* Inability to follow instructions
* Known kidney failure
* Heart failure with pitting oedema
* Thrombophlebitis
* Thromboembolic event during the previous three months
* Other surgery during the previous month
* Known malignancy
* Haemophilia; and pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Deep venous thrombosis (DVT) | Six weeks
  At 2 and 6 weeks postoperatively the number of participants with DVT will be assessed by compression duplex ultrasound (CDU)

SECONDARY OUTCOMES:
Functional outcome - muscular endurance tests (heel-rise) | Four years
  The functional outcome will be assessed at 26 and 52 weeks and 3-4 years postoperatively by validated muscular endurance test, i.e. heel rise test.
Patient-reported outcome - ATRS | Four years
  The patients' symptoms will be assessed using the reliable and valid score; the Achilles tendon Total Rupture Score (ATRS). 6, 12 months and 3-4 years postoperatively
Patient-reported outcome - EQ-5D | One year
  The patients' symptoms will be assessed using the reliable and valid score; EuroQol Group's questionnaire (EQ-5D).
Physical activity - PAS | Four years
  The patients' physical activity levels will be assessed a valid score; the Physical Activity scale (PAS). 6, 12 months and 3-4 years postoperatively
Patient-reported outcome - The Foot and Ankle Outcome Score (FAOS) | One year
  The patients' symptoms will be assessed using the reliable and valid score; The Foot and Ankle Outcome Score. FAOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Functioning sport and recreation (Sport(Rec), and foot and ankle-related Quality of Life (QOL). Each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. Assessed 6 and 12 months postoperatively
Patient-reported outcome - RAND 36 Health and Quality of Life questionnaire | One year
  The patients' symptoms will be assessed using the reliable and valid score; The RAND-36 Health and Quality of Life. The questionnaire is composed of 36 items, scored from 1 to 2,3, 5 or 6, some items are scored reversed. The score is divided in 8 subscales (dimensions) as the SF-36 questionnarie. The software recodes the points to a scale of 0 (worst) to 100 (best) for each subscale. Assessed at 6 and 12 months postoperatively
Patient-reported outcome - Tampa Scale of Kinesiophobia, Swedish version, TSK-SV | One year
  The patients' symptoms will be assessed using the reliable and valid score; The Tampa Scale of Kinesiophobia-SV. The scale comprises of 17 items and a total score is computed. 4 items are inverted and rescaled Before summation. Each item are scored from 1 (strongly disagree) to 4 (strongly agree). The total sum is between 17 to 68, where a score of more than 37 is defined as kinesiophobia. Assessed at 2 and 6 weeks and 6 and 12 months postoperatively
Plantar force loading | Six weeks
  Measured with mobile force sensors, insoles at 2 and 6 weeks postoperatively
Patient-reported diary - self-reported loading | Two weeks
  Estimation on daily self-reported loading on a VAS-scale, scored from 0 (non-weightbearing) to 100 (full weightbearing). Performed at home during the first 2 weeks postoperatively. The VAS scale is converted to percent (%) for analysis.
Patient-reported diary - pain ratings | Two weeks
  Pain ratings on a VAS-scale at home during the first week postoperatively. The patients are rating their pain from 0 (no pain) to 100 (worst imaginable pain) during activity and at rest.
Patient-reported diary - steps/day | Two weeks
  Measurement of number of steps taken each day with a valid pedometer at home during the first 2 weeks postoperatively
Calf circumference | Four years
  Measured with a tape measure at the thickest part of the calf in sitting position at 2 and 6 weeks and 6, 12 months and 3-4 years postoperatively
Ankle dorsiflexion | Six weeks
  Ankle range of motion in dorsiflexion, measured in sitting position with goniometer at 2 and 6 weeks postoperatively
Tendon length measurement | Four years
  Ultrasound measurement on Achilles tendon length, measured in centimeters, from the calcaneal bone to the gastrocnemius and the soleus muscles, with extended field-of-view images. Images taken at 2 and 6 weeks and 6 and 12 months and 3-4 years postoperatively
Tendon thickness measurement | One year
  Ultrasound measurement on Achilles tendon circumference (thickness), measured in cm2, with B-mode images. Images taken at 2 and 6 weeks and 6 and 12 months postoperatively
Muscle volume of the calf muscles | One year
  Ultrasound measurement on muscle volume of the calf muscles (gastrocnemius), measured in cm2, with extended field-of-view images. Images taken at 2 and 6 weeks and 6 and 12 months postoperatively
Thickness of the calf muscles | One year
  Ultrasound measurement on thickness of the calf muscle (soleus). Measured in centimeter, with B-mode images. Images taken at 2 and 6 weeks and 6 and 12 months postoperatively
Achilles Tendon resting angle (ATRA) | Four years
  A clinical measurement of indirect Tendon length with patient prone lying, measured with goniometer with arms parallell to fibula and MTP5, measured at 2 and 6 weeks and 6 and 12 months and 3-4 years postoperatively
3D gait analysis | 6 months
  Three-dimensional gait analysis, performed at 8 weeks and 6 months postoperatively, measurement of the quality of gait

OTHER OUTCOMES:
Tendon healing using microdialysis | Two weeks
  Microdialysis will be followed by quantification of markers for tendon repair
Time to surgery | Within 10 days
  Prognostic factor:
  Time to surgery , i.e. the time from ATR injury to start of the surgical procedure, will be calculated by using the time-point at which the patient sustained the injury as described in the patient journal, as well as the starting time point of the surgery as registered in the computerized operation report.
Surgeon sex | Surgery is performed within 10 days after injury
  Prognostic factor: All patients are operated on according to a standardized surgical protocol. and the surgeon on duty will perform the surgical repair and no specific surgeon can be selected by the patients. Unknown sex of the operating surgeon will be included as an additional exclusion criterion in the study.
Surgeon experience | Surgery is performed within 10 days after injury
  Prognostic factor: All patients are operated on according to a standardized surgical protocol. and the surgeon on duty will perform the surgical repair and no specific surgeon can be selected by the patients. The experienced group of surgeons will consist of specialists accredited with a specialist licence issued by The Swedish National Board of Health and Welfare. The less experienced group of surgeons will consist of residents.

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Ackermann, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska university Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Saarensilta A, Aufwerber S, Gravare Silbernagel K, Ackermann P. Early Tendon Morphology as a Biomarker of Long-term Patient Outcomes After Surgical Repair of Achilles Tendon Rupture: A Prospective Cohort Study. Orthop J Sports Med. 2023 Nov 6;11(11):23259671231205326. doi: 10.1177/23259671231205326. eCollection 2023 Nov. PMID 37941888
- [Derived] Chen J, Wang J, Hart DA, Zhou Z, Ackermann PW, Ahmed AS. Complement factor D regulates collagen type I expression and fibroblast migration to enhance human tendon repair and healing outcomes. Front Immunol. 2023 Sep 6;14:1225957. doi: 10.3389/fimmu.2023.1225957. eCollection 2023. PMID 37744351
- [Derived] Wu X, Chen J, Sun W, Hart DA, Ackermann PW, Ahmed AS. Network proteomic analysis identifies inter-alpha-trypsin inhibitor heavy chain 4 during early human Achilles tendon healing as a prognostic biomarker of good long-term outcomes. Front Immunol. 2023 Jul 6;14:1191536. doi: 10.3389/fimmu.2023.1191536. eCollection 2023. PMID 37483617
- [Derived] Aufwerber S, Silbernagel KG, Ackermann PW, Naili JE. Comparable Recovery and Compensatory Strategies in Heel-Rise Performance After a Surgically Repaired Acute Achilles Tendon Rupture: An In Vivo Kinematic Analysis Comparing Early Functional Mobilization and Standard Treatment. Am J Sports Med. 2022 Dec;50(14):3856-3865. doi: 10.1177/03635465221129284. Epub 2022 Nov 2. PMID 36322396
- [Derived] Chen J, Wang J, Hart DA, Ahmed AS, Ackermann PW. Complement factor D as a predictor of Achilles tendon healing and long-term patient outcomes. FASEB J. 2022 Jun;36(6):e22365. doi: 10.1096/fj.202200200RR. PMID 35596679
- [Derived] Aufwerber S, Edman G, Gravare Silbernagel K, Ackermann PW. Changes in Tendon Elongation and Muscle Atrophy Over Time After Achilles Tendon Rupture Repair: A Prospective Cohort Study on the Effects of Early Functional Mobilization. Am J Sports Med. 2020 Nov;48(13):3296-3305. doi: 10.1177/0363546520956677. Epub 2020 Sep 28. PMID 32986466
- [Derived] Aufwerber S, Heijne A, Edman G, Silbernagel KG, Ackermann PW. Does Early Functional Mobilization Affect Long-Term Outcomes After an Achilles Tendon Rupture? A Randomized Clinical Trial. Orthop J Sports Med. 2020 Mar 16;8(3):2325967120906522. doi: 10.1177/2325967120906522. eCollection 2020 Mar. PMID 32206673
- [Derived] Aufwerber S, Heijne A, Gravare Silbernagel K, Ackermann PW. High Plantar Force Loading After Achilles Tendon Rupture Repair With Early Functional Mobilization. Am J Sports Med. 2019 Mar;47(4):894-900. doi: 10.1177/0363546518824326. Epub 2019 Feb 11. PMID 30742483
- [Derived] Alim MA, Svedman S, Edman G, Ackermann PW. Procollagen markers in microdialysate can predict patient outcome after Achilles tendon rupture. BMJ Open Sport Exerc Med. 2016 Jun 10;2(1):e000114. doi: 10.1136/bmjsem-2016-000114. eCollection 2016. PMID 27900179

DOCUMENTS (1):
  • Study Protocol (2015-03-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT02318472/Prot_000.pdf